CLINICAL TRIAL: NCT00549341
Title: A Phase I, Single-dose, Double-blind, Placebo Controlled, Dose Escalation Study to Evaluate the Safety of PurTox for the Treatment of Adult Onset Spasmodic Torticollis/Cervical Dystonia and to Explore Dose-associated Efficacy
Brief Title: PurTox (Botulinum Toxin Type A) for the Treatment of Adult Onset Spasmodic Torticollis/Cervical Dystonia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT-ST-01
Record Dates: First submitted 2007-10-23; First posted 2007-10-25 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Spasmodic Torticollis
Keywords: Torticollis; Cervical Dystonia
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Mentor Purified Toxin, Botulinum Toxn Type A, Purified Neurotoxin
- 2 (Placebo Comparator)
  Interventions: Other: Physiologic saline

INTERVENTIONS:
Drug: Mentor Purified Toxin, Botulinum Toxn Type A, Purified Neurotoxin — 100U vials, doses ranged from 50U-200U, single injection.
  Arms: 1
Other: Physiologic saline — Single injection.
  Arms: 2

SUMMARY:
The safety and efficacy of Mentor Purified Toxin, Botulinum Toxin Type A, Purified Neurotoxin, injected intramuscularly into the neck, is being evaluated as a treatment for painful and non-painful spasmodic torticollis/cervical dystonia. It is hypothesized that treatment will decrease symptom severity and will not have any significant side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of torticollis with noticeable symptoms for at least 6 months
* Total TWSTRS score greater or equal to 20, TWSTRS severity score greater than or equal to 10 and TWSTRS Disability score greater than or equal to 3 (must meet all 3 criteria)

Exclusion Criteria:

* Diagnosis of isolated anterocollis
* Concurrent myopathic disease, myotonic dystrophy (or other form of muscular dystrophy), myasthenia gravis
* Currently receiving aminoglycoside antibiotic therapy, curare-like drugs, quinidine, succinylcholine, polymixins, anticholinesterases, magnesium sulfate, or lincosamides
* Any illness that is considered by the Investigator to make the subject an inappropriate candidate
* Cervical spine injury within 18 months or head and neck surgery within 6 months prior to screening
* Pre-existing dysphagia
* History of active autoimmune disease
* Exposure to botulinum toxin based pharmaceutical within 3 months prior to screening
* History of primary non-response or secondary resistance with prior exposure to botulinum based pharmaceuticals
* History of chemotherapy/radiation for malignant disease within 24 months
* Any investigational drug/device during the 30 days prior to screening

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-05; Primary Completion 2008-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Absence of significant drug related adverse effects | Post-injection

SECONDARY OUTCOMES:
Decrease in symptom severity (TWSTRS) | 30 days post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Austin, Study Director — Mentor Worldwide, LLC
Locations (1):
- Mentor Worldwide, LLC, Santa Barbara, California, United States